CLINICAL TRIAL: NCT06264193
Title: The Effects of Live High-train Low on EPO, VEGF, and Hematological Variables in Elite Rowers
Brief Title: The Impact of Hypoxia on the Biochemical and Morphological Parameters of Blood in Rowers.
Acronym: IHOBMPBR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Rowers LH-TL
Record Dates: First submitted 2024-01-10; First posted 2024-02-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2023-11

CONDITIONS: Hypoxia
Keywords: hypoxia; rowers; exercise; EPO; athletes; LH-TL
MeSH Terms: conditions — Hypoxia; Motor Activity

STUDY DESIGN:
Intervention Model Description: The hypoxic group included rowers participating in sports training and the LH-TL method, hypoxic rooms (FiO2=14.5%, corresponds to an altitude of 3000 meters). And the control group participating only in sports training and living in normoxic rooms, at the same sports camp.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxia (Experimental): live high-train low method was used
  Interventions: Other: hypoxia

INTERVENTIONS:
Other: hypoxia — The athletes were living in hypoxic rooms, and training was carried out on lowlands.

SUMMARY:
The response to hypoxia is very individual and epending on many aspects, such as the type of training, duration, intensity, or hypoxic stimulus, hypoxia affects the athlete in various ways. The results of this study have shown that 18 days of the LH-TL method does not significantly increase the level of EPO and VEGF in rowers. However, reticulocytes, immature red blood cells, have shown significant differences after 18-d LH-TL between groups. Further research should be carried out to investigate an optimal hypoxic dose and time, which will raise EPO, VEGF, and morphology variables.

DETAILED DESCRIPTION:
The Polish national rower team athletes, 13 males (ages 27,0±4,2 years), were randomly divided into two groups: 1) The hypoxic group (H) included 8 rowers participating in sports training and the LH-TL method, hypoxic rooms (FiO2=14.5%, corresponds to an altitude of 3000 meters). 2) The control group (C) presented 5 rowers participating only in sports training and living in normoxic rooms, at the same sports camp. Rowers were observed during the preparatory period. The hypoxic group lived and slept in hypoxic rooms, for at least 8-14 hours per day. During the camp, all rowers followed the same training schedule and diet.All participants' saturation and heart rate were measured daily, morning and evening, throughout the camp period. Venous blood samples were taken four times, at the beginning of the camp (Baseline), after 5 days, after 12 days, and after 18 days of the camp. Body composition parameters such as body mass index, body fat, and free fat mass were estimated using the bioelectrical impedance method of an analyzer Tanita BC 418 (Japan). Data analysis was performed using Statistica. The response to hypoxia is very individual. Depending on many aspects, such as the type of training, duration, intensity, or hypoxic stimulus, hypoxia affects the athlete in various ways. The results of this study have shown that the blood parameters did not increase significantly in the hypoxic group compared to the control group. However, reticulocytes, immature red blood cells, have shown significant differences after 18-d LH-TL between groups. Further research should be carried out to investigate an optimal hypoxic dose and time, which will raise EPO, VEGF, and morphology variables.

ELIGIBILITY:
Inclusion Criteria:

* member of national rower's teams, and sports camp participant.

Exclusion Criteria:

* negative symptoms of hypoxia, and/or injury.

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11-30 (Actual); Primary Completion 2014-12-21 (Actual); Study Completion 2014-12-21 (Actual)

PRIMARY OUTCOMES:
Erythropoietin (EPO) mlU/ml | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  immunoenzymatic assay methods using diagnostic kits
vascular endothelial growth factor (VEGF) mlU/ml | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  immunoenzymatic assay methods using diagnostic kits

SECONDARY OUTCOMES:
creatine kinase (CK) ng/ml | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  was determined using spectrophotometer analysis and diagnostic kits
Hs C-Reactive Protein (hsCRP) mg/L | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  was determined by immunoenzymatic assay methods using diagnostic kits
hemoglobin (Hb)g/dL | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  A professional accredited laboratory company determined the Hb level (Poland, ISO 9001:2008).
hematocrit (Htc)% | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  A professional accredited laboratory company determined the Htc level (Poland, ISO 9001:2008).
red blood cells (RBC)mln/mm3 | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  A professional accredited laboratory company determined the RBC level (Poland, ISO 9001:2008).
white blood cells (WBC)10 3/µL | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  A professional accredited laboratory company determined the WBC level (Poland, ISO 9001:2008).
reticulocytes (Ret)‰ | At the beginning of the camp (Baseline), after 5 days (T1), after 12 days (T2), and after 18 days (T3) of the camp.
  A professional accredited laboratory company determined the Ret level (Poland, ISO 9001:2008).
SpO2 - oxygen saturation (%) | every day, morning and evening, while sports camp
  was measured using a pulse oximeter (Tech-Med, ISO: 13485).
bpm - beats per minute(%) | every day, morning and evening, while sports camp
  was measured using a pulse oximeter (Tech-Med, ISO: 13485).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Kasperska, Principal Investigator — Poznań University of Physical Education, Faculty of Sport Sciences in Gorzów Wielkopolski, Poland;

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasperska A, Zembron-Lacny A. The effect of intermittent hypoxic exposure on erythropoietic response and hematological variables in elite athletes. Physiol Res. 2020 Apr 30;69(2):283-290. doi: 10.33549/physiolres.934316. Epub 2020 Mar 23. PMID 32199016
- [Background] Wilber RL. Application of altitude/hypoxic training by elite athletes. Med Sci Sports Exerc. 2007 Sep;39(9):1610-24. doi: 10.1249/mss.0b013e3180de49e6. PMID 17805095
- [Result] Czuba M, Fidos-Czuba O, Ploszczyca K, Zajac A, Langfort J. Comparison of the effect of intermittent hypoxic training vs. the live high, train low strategy on aerobic capacity and sports performance in cyclists in normoxia. Biol Sport. 2018 Mar;35(1):39-48. doi: 10.5114/biolsport.2018.70750. Epub 2017 Oct 11. PMID 30237660
- [Result] Ploszczyca K, Langfort J, Czuba M. The Effects of Altitude Training on Erythropoietic Response and Hematological Variables in Adult Athletes: A Narrative Review. Front Physiol. 2018 Apr 11;9:375. doi: 10.3389/fphys.2018.00375. eCollection 2018. PMID 29695978
- See also: Exercise and Training at Altitudes: Physiological Effects and Protocols — http://www.redalyc.org/pdf/562/56229795008.pdf